CLINICAL TRIAL: NCT03791047
Title: The Relationship Between Muscle Thickness and Dynamic Balance in Young and Older Adults
Brief Title: Evaluation of Muscle Thickness and Balance in Young and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GO 18/506
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy; Balance; Distorted
Keywords: Balance; Postural control; Muscle; Older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Balance analysis (Experimental): Sixty older subjects will be evaluated in this study. Muscle thickness and balance will be assessed by ultrasonography and Computerized Balance system respectively.
  Interventions: Other: Balance Analysis
- Control Group:Balance Analysis (Active Comparator): Sixty young subjects will be evaluated in this study. Muscle thickness and balance will be assessed by ultrasonography and Computerized Balance system respectively.
  Interventions: Other: Balance Analysis

INTERVENTIONS:
Other: Balance Analysis — Balance analysis is assessment method to estimate fall of risk and deterioration of postural control.

SUMMARY:
This study evaluates muscle thickness of trunk and lower limb and balance in young and older healthy adults. The participants will be evaluated muscle thickness for 14 different muscle and balance which evaluated by computerized force plate system.

DETAILED DESCRIPTION:
Aging had an adverse affect on musculoskeletal system and balance parameters. Decreased muscle strength or thickness negatively affect person's balance control. But there are no information in the literature about the relationships between muscle thickness and balance in healthy subjects. In addition to, it is not known which muscle responsible for balance. Therefore, this study will evaluate muscle thickness via ultrasonography and balance in young and older adults. Balance will be evaluated computerized Balance system. Muscle thickness for different 14 muscle ( diaphragm, transversus abdominis,multifidus, longissimus, quadratus lumborum, rectus abdominis, external and internal obliques, rectus femoris, vastus intermedius, vastus lateralis, tibialis anterior, gastrocnemius, soleus) will be evaluated by ultrasonography at the right side. Only diaphram muscle will be evaluated both right and left side.

ELIGIBILITY:
Inclusion Criteria For Young Adults:

* To be a volunteer to participate
* to be an aged 18-40 years old.

Inclusion Criteria For Older Adults:

* To be a volunteer to participate
* to be an aged 65-90 years old.

Exclusion Criteria:

* Walking with assist device
* Having a visual deficits
* Having an orthopedic problems that affect balance
* Having a neurological disorders
* Having a musculoskeletal disorders that affect balance
* Having an undergone orthopedic surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Limits of Stability | 15 minutes
  Limits of stability test evaluates dynamic balance of participants. Computerized balance system measured limits of stability for forward, backward, right and left side movements. It calculates the maximum distance a person can lean without losing balance. The unit of measure is centimeters. The higher value is indicated the better balance.

SECONDARY OUTCOMES:
Muscle thickness | 30 minutes
  Muscle thickness in millimeters by Ultrasound
Postural Sway | 15 minutes
  Postural sway in centimeters by computerized balance system
Fear of falling | 15 minutes
  Fear of Falling will be evaluated by Fall Efficacy Scale - International is a questionnaire that assesses fear of falling. The total scores range from 16 "absence of concern" to 64 "extreme concern.
Joint position sense | 15 minutes
  Knee joint position sense test will be evaluated using an isokinetic dynamometer. The testing included passive positioning performed by the assessor and active-repositioning performed by the participants. As the difference between the target degree and the degree is increased, the sense of position worsens.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozkal, Principal Investigator — Hacettepe University
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozkal O, Kara M, Topuz S, Kaymak B, Baki A, Ozcakar L. Assessment of core and lower limb muscles for static/dynamic balance in the older people: An ultrasonographic study. Age Ageing. 2019 Nov 1;48(6):881-887. doi: 10.1093/ageing/afz079. PMID 31268513